CLINICAL TRIAL: NCT01213459
Title: An Observational, Epidemiological Study on the Prevalence of Human Papillomavirus (HPV) Types in Women >= 15 Years of Age, in the Kingdom of Saudi Arabia
Brief Title: Study on the Prevalence of Human Papillomavirus Types in Women >= 15 Years of Age in the Kingdom of Saudi Arabia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 111336
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Infections, Papillomavirus; Cervical Cancer
Keywords: Human papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cervical samples

GROUPS / COHORTS (1):
- Cohort A: Women ≥15 years of age attending out-patient departments for routine cervical screening in the Kingdom of Saudi Arabia.
  Interventions: Procedure: Cervical samples; Other: Data collection

INTERVENTIONS:
Procedure: Cervical samples — Human papillomavirus detection and typing in cervical samples.
Other: Data collection — Questionnaire completion

SUMMARY:
This study aims to determine the prevalence of human papillomavirus (HPV) and to assess the HPV type distribution among women >= 15 years of age, attending routine gynaecological examination in the Kingdom of Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* Subjects/Subjects' parents or guardians, who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study,
* Women >=15 years of age attending a clinic for routine cervical screening,
* Written informed consent obtained from the subject and/or subject's parent/guardian.

Exclusion Criteria:

* Referral for abnormal cervical sample at the current visit,
* Abundant menstrual bleeding or vaginal discharge not allowing appropriate screening to be performed,
* No cervical sample provided,
* History of hysterectomy,
* Known diagnosis of immunosuppression, or patient on immunosuppressives,
* Pregnant female >=25 years of age.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women >=15 years of age attending out-patient departments of primary, secondary or tertiary care centers for routine cervical screening, in the Kingdom of Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2010-04; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of any human papillomavirus deoxyribo nucleic acid and of different types of human papillomavirus (including multiple infections) among women undergoing cervical screening. | At least 12 months from the date of subject enrolment

SECONDARY OUTCOMES:
Prevalence of any human papillomavirus deoxyribo nucleic acid and of different types of human papillomavirus (high risk and low risk) among women of different age strata undergoing cervical screening. | At least 12 months from the date of subject enrolment
Behavioural risk factors such as age at first marriage and age at first pregnancy (assessed through administration of a behavioural questionnaire). | At least 12 months from the date of subject enrolment
Level of awareness of human papillomavirus and its relation to transmission and to causation of cervical cancer. | At least 12 months from the date of subject enrolment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] AlObaid A, Al-Badawi IA, Al-Kadri H, Gopala K, Kandeil W, Quint W, Al-Aker M, DeAntonio R. Human papillomavirus prevalence and type distribution among women attending routine gynecological examinations in Saudi Arabia. BMC Infect Dis. 2014 Dec 14;14:643. doi: 10.1186/s12879-014-0643-8. PMID 25496614